CLINICAL TRIAL: NCT03026530
Title: Effect of Pulmonary Recruitment Maneuver (PRM) on Pain and Nausea After Laparoscopic Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Östergötland (Other)
Responsible Party: Principal Investigator, Ebba Kihlstedt Pasquier, Principal Investigator, Region Östergötland
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Region Östergötland
Record Dates: First submitted 2017-01-12; First posted 2017-01-20 (Estimated); Results first posted 2018-12-05 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Pain, Postoperative; Postoperative Nausea and Vomiting
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting | interventions — Ventilators, Mechanical

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Pulmonary recruitment maneuver (Experimental): Ventilator-piloted pulmonary recruitment maneuver at the end of laparoscopic bariatric surgery.
  Interventions: Procedure: Pulmonary recruitment maneuver; Procedure: Laparoscopic bariatric surgery; Device: Ventilator
- Control group (Active Comparator): Ordinary ventilation at the end of laparoscopic bariatric surgery.
  Interventions: Procedure: Laparoscopic bariatric surgery; Device: Ventilator

INTERVENTIONS:
Procedure: Pulmonary recruitment maneuver — The participants in the experimental arm receives 1 minute of ventilator-piloted pulmonary recruitment with positive inspiratory pressure set to 40 cm H2O, at the end of laparoscopic bariatric surgery.
  Arms: Pulmonary recruitment maneuver
Procedure: Laparoscopic bariatric surgery
Device: Ventilator

SUMMARY:
The purpose of this prospective, blinded, randomized clinical trial is to investigate whether a ventilator-piloted PRM at the end of laparoscopic bariatric surgery could reduce overall postoperative pain and nausea.

ELIGIBILITY:
Inclusion Criteria:

* elective laparoscopic bariatric surgery (LBS)
* American Society of Anaesthesiologists (ASA) physical status classification I-II (with the exception of body mass index over 35 kg/m2)
* written consent

Exclusion Criteria:

* conversion to open surgery
* complication, Clavien-Dindo grade ≥ II

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-11; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ebba Kihlstedt Pasquier, MD, Principal Investigator — Vrinnevi Hospital, Norrköping, Sweden; Ellen Andersson, MD, PhD, Study Chair — Vrinnevi Hospital, Norrköping, Sweden

REFERENCES:
- [Result] Pasquier EK, Andersson E. Pulmonary recruitment maneuver reduces pain after laparoscopic bariatric surgery: a randomized controlled clinical trial. Surg Obes Relat Dis. 2018 Mar;14(3):386-392. doi: 10.1016/j.soard.2017.11.017. Epub 2017 Nov 22. PMID 29290563

RESULTS

PARTICIPANT FLOW:
Groups:
- Pulmonary Recruitment Maneuver: Ventilator-piloted pulmonary recruitment maneuver at the end of laparoscopic bariatric surgery.
  Pulmonary recruitment maneuver: The participants in the experimental arm receives 1 minute of ventilator-piloted pulmonary recruitment with positive inspiratory pressure set to 40 cm H2O, at the end of laparoscopic bariatric surgery.
  Laparoscopic bariatric surgery
  Ventilator
- Control Group: Ordinary ventilation at the end of laparoscopic bariatric surgery.
  Laparoscopic bariatric surgery
  Ventilator
Period: Overall Study
Arm/Group | Pulmonary Recruitment Maneuver | Control Group
Started | 100 | 100
Completed | 79 | 71
Not Completed | 21 | 29
Not completed — Lost to Follow-up | 19 | 24
Not completed — Protocol Violation | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pulmonary Recruitment Maneuver | Control Group | Total
Number analyzed (Participants) | 79 | 71 | 150
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 47 [34 to 53] | 44 [32 to 51] | 46 [33 to 52]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 54 | 121
  Male | 12 | 17 | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Sweden | 79 | 71 | 150
BMI [Median (Inter-Quartile Range); unit: kg/m2] | 38 [36 to 42] | 38 [36 to 42] | 38 [36 to 42]

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pain
Description: A questionnaire with a numeric rating scale (NRS) is used to evaluate pain intensity at 4, 12, 24, 36 and 48 hours postoperatively to assess pain intensity. The scale includes even numbers from 0 to 10, where 0 signifies no pain, and 10 signifies the worst imaginable pain.
Time Frame: 4, 12, 24, 36 and 48 hours after surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Pulmonary Recruitment Maneuver | Control Group
Number analyzed (Participants) | 79 | 71
score on a scale
  4 hr | 3 [1 to 3] | 2 [1 to 4]
  12 hr | 2 [1 to 4] | 3 [1 to 4]
  24 hr | 2 [1 to 3] | 3 [2 to 5]
  36 hr | 2 [1 to 3] | 2 [1 to 4]
  48 hr | 1 [0 to 2] | 1 [0 to 2.75]

2. Secondary Outcome: Postoperative Nausea
Description: A questionnaire was used to evaluate nausea at 4, 12, 24, 36 and 48 hours postoperatively. The questionnaire involved a numeric rating scale (NRS) from 0 to 10, where 0 signified no nausea, and10 the worst imaginable nausea.
Time Frame: 4, 12, 24, 36 and 48 hours after surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Pulmonary Recruitment Maneuver | Control Group
Number analyzed (Participants) | 79 | 71
score on a scale
  4 hr | 1 [0 to 3] | 1 [0 to 3]
  NRS 12 hr | 1 [0 to 3] | 1 [0 to 2]
  24 hr | 0 [0 to 1] | 0 [0 to 1]
  36 hr | 0 [0 to 0] | 0 [0 to 1]
  48 hr | 0 [0 to 0] | 0 [0 to 1]

ADVERSE EVENTS:
Arm/Group | Pulmonary Recruitment Maneuver | Control Group
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 0/100 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No